CLINICAL TRIAL: NCT04632368
Title: Targeting the Health Care Provider (HCP) Burnout Crisis During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00106191
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-05

CONDITIONS: Burnout, Professional; Stress, Psychological
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Eligible participants, on enrollment in the study, would be randomly assigned to meditation intervention group vs control group. Control group will be offered intervention at the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation Intervention Arm (Active Comparator): TM, a mind-body intervention that can reduce sympathetic arousal and promote a state of relaxation and calm, will be offered to a randomized group of eligible HCPs ( N=40)providing care during COVID-19 pandemic.
  Interventions: Behavioral: Transcendental Meditation
- Treatment as usual(TAU) Control Arm (No Intervention): Control group consists of eligible HCPs who are randomized to control group(N=40) and would not receive any intervention. At the end of 3 month study period, control group participants would be eligible for TM training.

INTERVENTIONS:
Behavioral: Transcendental Meditation — TM, a mind-body intervention that can reduce sympathetic arousal and promote a state of relaxation and calm, will be offered to HCPs dealing with COVID-19 pandemic
  Arms: Transcendental Meditation Intervention Arm

SUMMARY:
This single blind, randomized, controlled trial (RCT) evaluates, a nonpharmacological intervention, TM (Transcendental Meditation) for improving burnout (, as measured by self-reporting (survey), physiologic, and neuro-functional imaging studies in health care providers (HCPs) when practiced over 3 months' time. The investigators define HCPs as any physician, physician trainee, nurse, physician assistant, nurse practitioner or respiratory therapist.

HCPs will be screened by a single-item stress scale and Columbia Suicide Severity Rating Scale (CSSRS) to understand their stress level and exclusion criteria respectively. The Global Severity Index of the Brief Symptom Inventory (BSI)-18 Global Severity score will be used as the primary outcome for pre- and post-TM training (baseline, 1 vs. 3 months). In addition, the investigators will evaluate physiological markers of stress and cardiovascular resiliency such as 1) changes (pre/post-treatment) in heart rate variability (HRV) through wearables, 2) Galvanic Skin Response (GSR) - changes in sweat gland activity that result from changes in an emotional state. fMRI will be performed by the Duke Brain Imaging and Analysis Center (BIAC) on a subset of participants to evaluate changes A specifically developed mobile app will aid data collection as well as reminders for providers to aid compliance for meditation

DETAILED DESCRIPTION:
OVERALL HYPOTHESIS: HCPs who learn and practice TM will demonstrate significantly improved symptoms of burnout within 3 months, as measured by self-report (survey), physiologic, and neuro-functional imaging studies.

SPECIFIC AIM 1: To conduct a single-blind, randomized, controlled trial (RCT) of TM (N=40) vs. Control (CTL, N=40) in frontline HCPs. HCPs will be screened by a single-item stress scale and Columbia Suicide Severity Rating Scale (CSSRS). The Global Severity Index of the Brief Symptom Inventory (BSI)-18 Global Severity score will be used as the primary outcome for pre- and post-TM training (baseline, 1 vs. 3 months). SPECIFIC AIM 2: Evaluate changes (pre/post-treatment) in heart rate variability (HRV), a physiological measure of stress, and overall cardiovascular resilience) in response to TM practice versus CTL. Participants will be asked to wear an Apple Watch throughout trial participation to assess changes in resting HRV during meditative practice. Galvanic Skin Response (GSR) refers to the changes in sweat gland activity that result from changes in an emotional state. A portable GSR device (e-Sense Skin Response) will be used to evaluate GSR score (baseline and 3 months). fMRI (N=20 for each group) will be performed by the Duke Brain Imaging and Analysis Center (BIAC).

fMRI Protocol: The first 20 eligible (exclusion criteria: pregnancy, claustrophobia, reluctance to participate) patients from each group will be randomly assigned to get fMRI at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

HCPs including physicians, trainee physicians, nurses, nurse practitioners, Physician Assistants, and respiratory therapists providing patient care during the COVID-19 pandemic.

* A single-item stress scale will be used as a screen for eligibility; a minimum score of 6 on a 10-point response scale will be needed to meet inclusion criteria
* Subjects who have at least a 5% increase from baseline in heart rate after exposure to a personalized stressful script OR at least a 33% increase in skin conductance after exposure to the script
* Willingness to address burnout symptoms by non-pharmacological means
* All subjects must provide Informed Consent prior to enrollment in the study.
* Willingness to wear the provided Apple Watch for the data collection process

Exclusion Criteria:

* Antipsychotic medications or beta-blockers
* Current suicidal or homicidal ideation (suicidal ideation as screened by C-SSRI survey pre-enrollment)
* Previous instruction in TM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
change in self reported Stress symptoms | Baseline, 1 month, 3 months
  Changes in brief symptom inventory as evaluated by BSI 18

SECONDARY OUTCOMES:
Change in self reported resilience | Baseline, 1 month, 3 months
  These will include secondary outcomes as measured by the Connor Davidson Resilience Scale-25 (CD-RISC).
Change in symptoms of depression | Baseline, 1 month, 3 months
  Change in symptoms of depression will be measured by PHQ 9 scale
Change in insomnia symptoms | Baseline, 1 month, 3 months
  Change in insomnia symptoms as measured by Insomnia severity Index(ISI)
Change in anxiety symptoms | Baseline, 1 month, 3 months
  Change in anxiety symptoms as measured by GAD-7
Change in psychological distress | Baseline, 1 month, 3 months
  change in psychological distress as measured by the Global Severity Index of the Brief Symptom Inventory (BSI)-18 questionnaire.
Change in self reported burnout symptoms | Time Frame: Baseline, 1 month, 3 months
  Change in burnout symptoms in HCPs as measured by Maslach Burnout Inventory( MBI)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University health system, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi SP, Wong AI, Brucker A, Ardito TA, Chow SC, Vaishnavi S, Lee PJ. Efficacy of Transcendental Meditation to Reduce Stress Among Health Care Workers: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231917. doi: 10.1001/jamanetworkopen.2022.31917. PMID 36121655